CLINICAL TRIAL: NCT00002903
Title: PHASE II TRIAL WITH DOCETAXEL IN PATIENTS WITH RELAPSING GERM CELL CANCER
Brief Title: Docetaxel in Treating Patients With Recurrent or Refractory Germ Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16945T; EORTC-16945T
Record Dates: First submitted 1999-11-01; First posted 2004-05-13 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Extragonadal Germ Cell Tumor; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; testicular seminoma; recurrent ovarian germ cell tumor; extragonadal germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of docetaxel in treating patients with recurrent or refractory germ cell cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether partial or complete responses can be achieved with docetaxel (TXT) in patients with recurrent or refractory disseminated germ cell cancer previously treated with standard-dose chemotherapy. II. Assess the probability of actual response warranting further evaluation of the therapeutic effectiveness of TXT in the case that partial or complete tumor responses are achieved in this patient population. III. Characterize further the toxic effects of TXT in these patients.

OUTLINE: Patients receive intravenous docetaxel over 1 hour every 3 weeks until disease progression, unacceptable toxicity, or at least 3 courses beyond documentation of complete response. Patients may receive concurrent radiotherapy provided not all indicator lesions are included in irradiated field. Resection of residual mature teratoma is allowed no sooner than 8 weeks after therapy provided tumor markers are normalized for at least 4 weeks.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed extragonadal and gonadal germ cell tumor Seminoma and nonseminoma eligible Recurrent or refractory disease despite adequate first-line cisplatin- or carboplatin-based chemotherapy and not amenable to surgery and/or curative radiotherapy Relapse after disease-free interval of 1 or more years ineligible Measurable or evaluable disease with documented progression within 2 months prior to entry Elevated beta human chorionic gonadotropin and alpha-fetoprotein considered evaluable if no other evaluable lesion and provided marker(s): Increased since end of last treatment At least 10 times upper limit of normal unless due to tumor lysis Rising on 3 successive occasions at least 2-3 days apart If no tumor markers available, cytology or histology should be obtained No inadequately treated CNS metastases No pleural or pericardial effusion and/or ascites

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute granulocyte count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.25 times normal AST/ALT no greater than 3 times normal Alkaline phosphatase no greater than 2.5 times normal Renal: Creatinine no greater than 1.6 mg/dL Creatinine clearance at least 60 mL/min if creatinine borderline (1.1-1.6 mg/dL) Other: No active infection No severe malnutrition No pre-existing grade 2 or worse neurotoxicity No pre-existing edema No senility or psychosis No other expected difficulties for follow-up including geographic considerations No other malignancy except: Second testicular primary tumor Treated basocellular and planocellular skin carcinoma Adequately treated carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior high dose chemotherapy with or without stem cell transplant At least 3 weeks since chemotherapy and past WBC and platelet nadirs Endocrine therapy: Not specified Radiotherapy: Not amenable to curative radiotherapy At least 3 weeks since radiotherapy and recovered Surgery: Not amenable to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1995-07

CONTACTS AND LOCATIONS:
Overall Officials: Emma Geertruida Elisabeth De Vries, MD, PhD, Study Chair — University Medical Center Groningen
Locations (49):
- Ludwig Boltzmann - Institute for Applied Cancer Research, Vienna, Austria
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital - University Hospital of Copenhagen, Herlev
- France (14):
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Curie - Section Medicale, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Martin Luther Universitaet, Halle
  - Universitats-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
- University of Ioannina, Ioannina, Greece
- Israel (2):
  - Rambam Medical Center, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Italy (5):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - San Raffaele Hospital, Rome
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- Netherlands (5):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Switzerland (5):
  - University Hospital, Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern, Bern
  - Clinique De Genolier, Genolier
  - Kantonsspital - Saint Gallen, Sankt Gallen
- United Kingdom (4):
  - Royal Marsden NHS Trust, London, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland